CLINICAL TRIAL: NCT00089089
Title: Phase I Study of Prolonged Low Dose Decitabine (5-Aza-Deoxycytidine, NSC #127716) in Patients With Biopsiable Advanced Cancers Refractory to Standard Therapy
Brief Title: Decitabine in Treating Patients With Advanced Refractory Solid Tumors or Lymphomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03096; 2004-0040; U01CA062461 (NIH)
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Hematopoietic/Lymphoid Cancer; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Decitabine

ARMS (1):
- Treatment (decitabine) (Experimental): Patients receive decitabine IV over 1 hour on days 1-5 or on days 1-5 and 8-12. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Cohorts of 6 patients receive escalating doses of decitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.
  Interventions: Drug: decitabine; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: decitabine — Given IV
  Other Names: 5-aza-dCyd; 5AZA; DAC
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of decitabine in treating patients with metastatic or unresectable refractory solid tumors or lymphomas. Drugs used in chemotherapy, such as decitabine, work in different ways to stop cancer cells from dividing so they stop growing or die

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose of single agent decitabine and its toxicity using this schedule in this population of patients with solid tumors or lymphomas.

II. Definition of the dose at which tumor DNA demethylation is optimum. III. Definition of the dose at which peripheral blood mononuclear cell (PBMN) demethylation is optimal.

IV. Definition of decitabine pharmacokinetics and correlation of plasma concentrations with hypomethylation effects.

SECONDARY OBJECTIVES:

I. Preliminary assessment of decitabine efficacy (objective response).

OUTLINE: This is a dose-escalation study.

Patients receive decitabine IV over 1 hour on days 1-5 or on days 1-5 and 8-12. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 6 patients receive escalating doses of decitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed malignancy (solid tumor or lymphoma) that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* Patients must have had >= 1 prior chemotherapy regimen; there is no maximum allowable number of prior regimens, provided all other eligibility criteria are met
* Patients must be >= 6 weeks beyond treatment with a nitrosourea or mitomycin-C, >= 4 weeks beyond other chemotherapy or radiotherapy, and must have recovered to =< grade 1 toxicity for any treatment-limiting toxicity of prior therapy; (Exception: patients may have received palliative low dose radiotherapy to the limbs 1-4 weeks before this therapy, provided pelvis, ribs, sternum, scapulae, vertebrae or skull were not included in the radiotherapy field)
* ECOG performance status =< 2 (Karnofsky >= 60%); (Exception: Patients with brain metastases must be ECOG performance status 0-1)
* Leukocytes >= 3,000/μL
* Absolute neutrophil count >= 1,500/μL
* Platelets >= 140,000/μL
* Total bilirubin =< 1.0 mg/dL
* AST(SGOT)/ALT(SGPT) =< 1.5 X institutional upper limit of normal
* Creatinine (serum) =< 1.5 mg/dL
* PT within institutional guideline for biopsy procedure (=< to 16 seconds)
* The effects of decitabine on the developing human fetus are unknown; for this reason and because chemotherapy agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document, including consent for the required tumor biopsy, blood and pharmacokinetics studies
* Tumor accessible for repeat biopsy

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered to =< grade 1 treatment-limiting toxicity levels for adverse events due to agents administered more than 4 weeks earlier; (Exception: patients may have received palliative low dose radiotherapy to the limbs 1-4 weeks before this therapy provided pelvis, ribs, sternum, scapulae, vertebrae or skull were not included in the radiotherapy field)
* Patients who have had surgery within 2 weeks prior to entering the study
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases to whom any of the following apply:

  * Have not received prior cranial irradiation
  * Are requiring > 8 mg dexamethasone per day (or equivalent other steroid) to maintain an ECOG performance status =< 1
  * Have had a seizure (focal or generalized) in the last 3 weeks
  * If steroids required to maintain an ECOG performance status =< 1 have increased in the past 2 weeks
  * Take enzyme-inducing anti-convulsants
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to decitabine
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, potentially life threatening cardiac arrhythmia, systolic BP < 90 mmHg or > 160 mmHg, diastolic BP < 50 mmHg or > 110 mmHg, psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because decitabine is an antimetabolite with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with decitabine, breastfeeding should be discontinued if the mother is treated with decitabine
* Because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, patients known to be HIV-positive and receiving anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with decitabine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2004-09; Primary Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Phase II dose will be defined as the lowest dose at or below the maximum tolerated dose (MTD; based on dose limiting toxicity) consistent with a plateau reduction in DNA methylation in target tumor tissue | 4 weeks
Tumor demethylation response, measured by percent change in DNA methylation using the ALU assay | Baseline to day 12 course 1
  Analysis of variance with Fisher's protected least significant difference to group dose levels that elicit consistent demethylation response will be used.
Adequacy of peripheral blood mononuclear cell DNA methylation as a surrogate for tumor DNA methylation, measured by effect of dose on reduction in DNA methylation in peripheral blood mononuclear cells | Day 12 course 1
Pharmacokinetic parameters, including Cmax, Tmax, AUC, t ½ α, t ½ β, Vd, and clearance | Days 1 and 5 of course 1

SECONDARY OUTCOMES:
Response using RECIST | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: David Stewart, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States